CLINICAL TRIAL: NCT01011309
Title: A Phase 2, Randomized, Open-Label, Controlled Study to Evaluate the Efficacy, Safety, and Immunogenicity of the LEISH-F2 + MPL-SE Vaccine in the Treatment of Patients With Cutaneous Leishmaniasis
Brief Title: A Study of the Efficacy and Safety of the LEISH-F2 + MPL-SE Vaccine for Treatment of Cutaneous Leishmaniasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Access to Advanced Health Institute (AAHI) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDRI-LCVTC-202
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Results first posted 2013-11-18 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-11

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Leishmaniasis; vaccine; immunotherapy
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis | interventions — Antimony Sodium Gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LEISH-F2 + MPL-SE vaccine (Experimental): Recombinant three antigen Leishmania polyprotein + MPL-SE adjuvant
  Interventions: Biological: LEISH-F2 + MPL-SE
- Sodium stibogluconate (SSG) (Active Comparator): 20 mg/kg/day IV for 20 days
  Interventions: Drug: Sodium stibogluconate

INTERVENTIONS:
Biological: LEISH-F2 + MPL-SE — 10 μg LEISH-F2 + 25 μg MPL-SE on Days 0, 28 and 56
  Other Names: There are no other names for the vaccine.
  Arms: LEISH-F2 + MPL-SE vaccine
Drug: Sodium stibogluconate — 20 mg/kg/day IV daily for 20 days
  Other Names: Marfan SSG
  Arms: Sodium stibogluconate (SSG)

SUMMARY:
The purpose of this study is to determine the efficacy, safety, and immunogenicity of an investigational vaccine being developed for the treatment of leishmaniasis, including cutaneous leishmaniasis (CL). The vaccine, identified as LEISH-F2 + MPL-SE, consists of a Leishmania protein (LEISH-F2) together with an adjuvant MPL-SE.

DETAILED DESCRIPTION:
A phase 2, randomized, open-label, controlled study to evaluate the efficacy, safety, and immunogenicity of the vaccine administered three times (10 μg LEISH-F2 + 25 μg MPL-SE on Days 0, 28 and 56) in the treatment of adults and adolescents with CL compared to treatment with standard chemotherapy (20 mg/kg/day sodium stibogluconate for 20 days). The proportion cured in each group will be determined using clinical criteria.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 12 years and < 70 years of age. In the first stage of the study, only patients aged ≥ 18 years and < 70 years will be enrolled. In the second stage, enrollment will also include adolescent patients aged ≥ 12 - < 18 years.
* Must have a clinical diagnosis of cutaneous leishmaniasis confirmed by positive identification of Leishmania parasite and identification of L. peruviana by PCR.
* Lesions must be clear of any superinfection prior to enrollment.
* Female patients of childbearing age must have a negative serum pregnancy test at screening, a negative urine pregnancy test within 24 hours before the first vaccination or initiation of chemotherapy, must not be breast-feeding, and are required to use adequate contraception through Day 84 of the study. These precautions are necessary due to unknown effects that LEISH-F2 + MPL SE, sodium stibogluconate might have in a fetus or newborn infant.
* The following laboratory blood tests must have values within the normal ranges at screening: sodium, potassium, urea, total bilirubin, ALT, AST, glucose, creatinine, alkaline phosphatase, total WBC count and platelet count. Hemoglobin may exceed the ULN since patients reside in the Andes at very high altitude (up to 20 g/dL)
* The following serology tests must be negative at screening: HIV-1/2, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody. All patients (or their parents) will receive HIV-related counseling prior to testing. Patients with positive HIV test results will be referred for counseling and treatment as appropriate.
* Potential study patients (or their guardians) must give written informed consent, be willing to be housed in Lima for a minimum of 20 days and up to 63 days, able to attend all required follow-up visits, have a permanent address, and be reachable by study site personnel.

Exclusion Criteria:

* Infection with species other than L.peruviana as confirmed by PCR.
* Presence of eleven or more active cutaneous leishmaniasis lesions.
* The diameter of the ulcerated area of any single lesion is >60 mm.
* Presence of lesions with superinfection at time of enrollment.
* History of mucocutaneous leishmaniasis or diagnosis of mucocutaneous leishmaniasis at screening.
* History of previous exposure to Leishmania vaccines.
* Known use of injected or oral corticosteroids within 6 weeks prior to the first vaccination or initiation of chemotherapy.
* Participation in another experimental protocol or receipt of any investigational products within 30 days prior to the first vaccination or initiation of chemotherapy.
* History of autoimmune disease or other causes of immunosuppressive states.
* History or evidence of any acute or chronic illness that, in the opinion of the study clinician, may interfere with the evaluation of the safety or the immunogenicity of the vaccine. (Patients presenting with concomitant illness will be referred for standard clinical care).
* History of use of any medication that, in the opinion of the study clinician, may interfere with the evaluation of the safety or the immunogenicity of the vaccine.
* History of significant psychiatric illness.
* Drug addiction including alcohol abuse.
* Patients with a history of previous anaphylaxis, severe allergic reaction to vaccines or unknown allergens, or allergic reaction to eggs.
* Patients who are unlikely to cooperate with the requirements of the study protocol.
* ECG with evidence of ventricular arrythmias ≥ 4 extra systoles per minute.
* Known allergy or contraindication to chemotherapy (e.g., known reaction to pentavalent antimonials, cardiopathy, myocarditis).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-10; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franco Piazza, MD, MPH, Study Director — Access to Advanced Health Institute (AAHI)
Locations (1):
- Instituto de Medicina Tropical"Alexander von Humboldt", Lima, Peru

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with CL were actively recruited from Andean mountain regions endemic for transmission of Leishmania peruviana. Patients were treated in a medical clinic at the Instituto de Medicina Tropical 'Alexander von Humboldt', Universidad Peruana Cayetano Heredia, Lima, Peru.
Pre-assignment Details: All eligible patients were randomized to treatment groups. One patient was mistakenly randomized (ineligible) and was not treated.
Groups:
- Immunotherapy v1.4/1.5: 10 mcg LEISH-F2 antigen + 25 mcg MPL-SE adjuvant given as three subcutaneous injections on Days 0, 28, and 56.
- Immunotherapy v1.6: 10 mcg LEISH-F2 antigen + 25 mcg MPL-SE adjuvant given as three subcutaneous injections on Days 0, 14, and 28.
- Chemotherapy: Sodium stibogluconate (SSG) given 20 mg/kg/day IV for 20 days.
Period: Overall Study
Arm/Group | Immunotherapy v1.4/1.5 | Immunotherapy v1.6 | Chemotherapy
Started | 14 | 10 | 21
Completed | 12 | 7 | 16
Not Completed | 2 | 3 | 5
Not completed — Adverse Event | 2 | 1 | 2
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immunotherapy v1.4/1.5 | Immunotherapy v1.6 | Chemotherapy | Total
Number analyzed (Participants) | 14 | 10 | 21 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 10 | 20 | 44
  >=65 years | 0 | 0 | 1 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 38.3 (14.2) | 32.7 (6.8) | 40.2 (16.0) | 38.0 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 8 | 18
  Male | 9 | 5 | 13 | 27
Region of Enrollment [Number; unit: participants]
  Peru | 14 | 10 | 21 | 45

OUTCOME MEASURES:

1. Primary Outcome: Date of Clinical Cure
Description: Efficacy of immunotherapy with the LEISH-F2 + MPL-SE vaccine was compared to the efficacy of chemotherapy with sodium stibogluconate in the treatment of CL. Efficacy is measured by the date of clinical cure.
Time Frame: Day 84
Population: Per-protocol population: All patients who received all three study injections if in the immunotherapy groups or at least 15 injections of SSG if in the chemotherapy group, and completed the Day 56 visit (Immunotherapy v1.6), the Day 84 visit (Immunotherapy v1.4/1.5), or the Day 56 or Day 84 visit (Chemotherapy group).
Measure: Number; unit: participants
Arm/Group | Immunotherapy v1.4/1.5 | Immunotherapy v1.6 | Chemotherapy
Number analyzed (Participants) | 12 | 7 | 16
participants
  Clinical cure by Day 84 without rescue treatment | 2 | 2 | 15
  Clinical cure by Day 84 with rescue treatment | 10 | 5 | 1

2. Primary Outcome: Adverse Events of Grade 1 Severity or Higher Occurring in ≥ 3 Patients During Active Treatment Phase of the Study.
Description: Safety of immunotherapy with the vaccine was compared to the safety of chemotherapy with sodium stibogluconate. All adverse events are listed regardless of relatedness.
Time Frame: Day 0 through Day 84
Population: Safety population: All patients who received at least one study injection.
Measure: Number; unit: participants
Arm/Group | Immunotherapy v1.4/1.5 | Immunotherapy v1.6 | Chemotherapy
Number analyzed (Participants) | 14 | 10 | 21
participants
  Injection site erythema | 10 | 9 | 0
  Injection site induration | 8 | 10 | 0
  Injection site pain | 8 | 10 | 0
  Superinfection bacterial | 4 | 0 | 0
  ALT increased | 8 | 4 | 10
  Alkaline phosphatase increased | 5 | 1 | 1
  Total bilirubin increased | 4 | 1 | 3
  Hemoglobin decreased | 3 | 0 | 7
  WBC decreased | 4 | 1 | 10
  Headache | 3 | 3 | 5
  Nausea | 0 | 0 | 3

3. Secondary Outcome: IgG Antibodies and T-cell Cytokine Responses (IFN-g and IL-10)
Description: Immunogenicity of the vaccine was evaluated by measuring IgG antibody and T-cell responses to the LEISH-F2 protein and soluble Leishmania antigen (SLA). IgG antibodies were measured by ELISA and T-cell cytokine responses (IFN-g and IL-10) were measured by Luminex. Data is presented as median Post:Pre ratios comparing Days 56/84 or 168 to baseline at Day 0.
Time Frame: Days 0, 56 or 84, and 168
Population: Per-protocol population: patients who received all three study injections (immunotherapy groups) or at least 15 SSG injections (chemotherapy group) and completed the Day 84 or Day 56 visit.
Measure: Median (Full Range); unit: Relative ELISA Units
Arm/Group | Immunotherapy v1.4/1.5 | Immunotherapy v1.6 | Chemotherapy
Number analyzed (Participants) | 12 | 7 | 16
Relative ELISA Units
  IgG antibody to LEISH-F2 - Day 56 | NA [NA to NA] — Immunogenicity not measured at Day 56 in Immunotherapy v1.4/1.5. | 84.56 [40.99 to 409.8] | 2.004 [0.392 to 37.02]
  IgG antibody to LEISH-F2 - Day 84 | 76.72 [31.19 to 577.1] | NA [NA to NA] — Immunogenicity not measured at Day 84 in Immunotherapy v1.6. | 0.662 [0.176 to 104.3]
  IgG antibody to LEISH-F2 - Day 168 | 23.93 [6.74 to 159.6] | 10.26 [9.11 to 80.75] | 0.74 [0.24 to 1.29]
  IgG antibody to SLA - Day 56 | NA [NA to NA] — Immunogenicity not measured at Day 56 in Immunotherapy v1.4/1.5. | 1.36 [0.46 to 3.14] | 0.59 [0.17 to 1.44]
  IgG antibody to SLA - Day 84 | 1.6 [0.84 to 4.43] | NA [NA to NA] — Immunogenicity not measured at Day 84 in Immunotherapy v1.6. | 0.54 [0.11 to 3.12]
  IgG antibody to SLA - Day 168 | 0.63 [0.15 to 2.88] | 0.95 [0.08 to 1.19] | 0.33 [0.05 to 0.89]
  IFN-g response to LEISH-F2 - Day 56 | NA [NA to NA] — Immunogenicity not measured at Day 56 in Immunotherapy v1.4/1.5. | 4.97 [0.354 to 38.36] | 1.09 [0.003 to 34.71]
  IFN-g response to LEISH-F2 - Day 84 | 0.92 [0.042 to 19.13] | NA [NA to NA] — Immunogenicity not measured at Day 84 in Immunotherapy v1.6. | 1.333 [0.073 to 296.8]
  IFN-g response to LEISH-F2 - Day 168 | 1.00 [0.04 to 4.76] | 2.06 [0.41 to 11.3] | 0.82 [0.15 to 19.6]
  IFN-g response to SLA - Day 56 | NA [NA to NA] — Immunogenicity not measured at Day 56 in Immunotherapy v1.4/1.5. | 0.87 [0.09 to 6.1] | 0.84 [0.01 to 75.3]
  IFN-g response to SLA - Day 84 | 0.27 [0.02 to 39.7] | NA [NA to NA] — Immunogenicity not measured at Day 84 in Immunotherapy v1.6. | 0.89 [0.09 to 29.8]
  IFN-g response to SLA - Day 168 | 0.2 [0.01 to 76.5] | 0.31 [0 to 2.5] | 0.69 [0.05 to 3.94]
  IL-10 response to LEISH-F2 - Day 56 | NA [NA to NA] — Immunogenicity not measured at Day 56 in Immunotherapy v1.4/1.5. | 3.16 [0.4 to 12.8] | 1.22 [0.06 to 8.73]
  IL-10 response to LEISH-F2 - Day 84 | 1.44 [0.57 to 47.2] | NA [NA to NA] — Immunogenicity not measured at Day 84 in Immunotherapy v1.6. | 1.17 [0.06 to 18.9]
  IL-10 response to LEISH-F2 - Day 168 | 2.19 [0.16 to 27.5] | 0.9 [0.44 to 3.48] | 1.03 [0.08 to 4.91]
  IL-10 response to SLA - Day 56 | NA [NA to NA] — Immunogenicity not measured at Day 56 in Immunotherapy v1.4/1.5. | 1.02 [0.64 to 2.68] | 0.69 [0.03 to 7.44]
  IL-10 response to SLA - Day 84 | 0.63 [0.15 to 25.2] | NA [NA to NA] — Immunogenicity not measured at Day 84 in Immunotherapy v1.6. | 0.92 [0.04 to 9.85]
  IL-10 response to SLA - Day 168 | 0.952 [0.062 to 308.9] | 0.565 [0.294 to 1.068] | 0.763 [0.177 to 3.737]

ADVERSE EVENTS:
Time Frame: Day 0 through Day 336.
Description: All SAEs are listed regardless of relatedness. Other adverse events listed are considered possibly, probably, or definitely related to study vaccination or chemotherapy.
Arm/Group | Immunotherapy v1.4/1.5 | Immunotherapy v1.6 | Chemotherapy
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/10 | 1/21
Other Adverse Events (participants affected / at risk) | 13/14 | 10/10 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunotherapy v1.4/1.5 (N=14) | Immunotherapy v1.6 (N=10) | Chemotherapy (N=21)
Hospitalization due to Antimonial Toxicity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Unrelated to vaccination. Headache, nausea, vomiting, abdominal pain and oral discomfort. Lab tests: potassium 2.1mmol/L (Grade 4); AST 66U/L (Grade 1); ALT 35U/L (Grade 1); WBC 3900/mm3 (Grade 1); hgb 10.9g/dL (Grade 1); platelets 65K/mm3 (Grade 2).
Hospitalization due to Grade 3 Cellulitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Unrelated to study vaccination. First and second degree burns caused by spilled hot water on left thigh and knee. The subject was treated immediately; pain was well controlled and subsided within 24 hours.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Immunotherapy v1.4/1.5 (N=14) | Immunotherapy v1.6 (N=10) | Chemotherapy (N=21)
ALT increased (Investigations) | 8 (8) | 3 (3) | 9 (10)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (4) | 1 (1) | 3 (3)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 4 (4)
Blood sodium increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (3) | 0 (0) | 7 (7)
Headache (Nervous system disorders) | 1 (1) | 2 (4) | 5 (5)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Injection site erythema (General disorders) | 10 (13) | 9 (21) | 0/0 (0)
Injection site induration (General disorders) | 8 (9) | 10 (21) | 0/0 (0)
Injection site pain (General disorders) | 8 (12) | 10 (25) | 0/0 (0)
Malaise (General disorders) | 0 (0) | 2 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Superinfection bacterial (Investigations) | 1 (1) | 0 (0) | 0 (0)
WBC decreased (Investigations) | 2 (2) | 0 (0) | 10 (10)

LIMITATIONS AND CAVEATS:
A total of 150 patients was planned, including age de-escalation to adolescents after the first 60 adults enrolled. Owing to slow recruitment and insufficient evidence of efficacy in the immunotherapy group, enrollment was closed early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
IDRI encourages publication in peer-reviewed medical journals and will not unduly withhold permission to publish. However, all proposed publications, papers, abstracts or written materials related to the study or an outline of any oral presentation, shall be submitted to and coordinated by IDRI to assure that no proprietary information is presented and that authorship is fairly represented.